CLINICAL TRIAL: NCT01245790
Title: An Open-label, Phase I Study to Assess the Pharmacokinetics of R406 in Subjects With Renal Impairment Compared to Healthy Subjects Following Administration of a Single Dose of Fostamatinib 150 mg
Brief Title: A Study of Fostamatinib in Subjects With Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00009
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis; Renal Impairment
Keywords: Phase 1; healthy volunteers; volunteers with renal impairment; pharmacokinetics; Rheumatoid arthritis; RA; fostamatinib; Patients
MeSH Terms: conditions — Arthritis, Rheumatoid; Renal Insufficiency | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Healthy subjects (Stage 1)
  Interventions: Drug: fostamatinib
- 2 (Experimental): Mild renal impairment (Stage 2)
  Interventions: Drug: fostamatinib
- 3 (Experimental): Moderate renal impairment (Stage 2)
  Interventions: Drug: fostamatinib
- 4 (Experimental): Severe renal impairment (Stage 2)
  Interventions: Drug: fostamatinib
- 5 (Experimental): End stage renal disease (Stage 1)
  Interventions: Drug: fostamatinib

INTERVENTIONS:
Drug: fostamatinib — Oral tablets, single dose

SUMMARY:
A 2 stage study to evaluate the amount of fostamatinib in the blood and urine in subjects with impaired kidney (renal) function compared with healthy volunteers with normal renal function. Stage 1 will include healthy subjects and subjects with end stage renal disease, while Stage, 2 may include subjects with mild, moderate and/or severe renal impairment dependent on the outcome of Stage 1. The study will also evaluate safety and tolerability in subjects with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (non child bearing potential) greater than or equal to 18 years of age with suitable veins for cannulation or repeated venipuncture and with a weight of at least 50 kg (110 lbs) and body mass index (BMI) between 18 and 40 kg/m2, inclusive
* Stable renal impairment with following creatinine clearance (CLCR): Stage 1 - End Stage Renal Disease (ESRD) < 15 mL/min (requiring dialysis); Stage 2 - Mild renal impairment ≥ 50 to < 80 mL/min; Moderate renal impairment ≥ 30 to <50 mL/min; and severe renal impairment 15 to < 30 mL/min
* Healthy subjects with normal renal function must have good health based on medical history, physical examination , echocardiogram and clinical laboratory evaluations including creatinine clearance >80 ml/min"
* Negative screen for Human Immunodeficiency Virus and negative results for serum hepatitis B surface antigen and hepatitis C antibody

Exclusion Criteria:

* Subjects who have received any medications known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration
* Absolute neutrophil count less than 1600/mm3 or 1.6 x 109 L.
* Healthy subjects only: Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration
* Subjects with a history of multiple drug allergies or with a known allergy to the drug class of fostamatinib
* In the opinion of the Investigator, any evidence of additional severe or uncontrolled systemic disease (eg, currently unstable or uncompensated hepatic, cardiovascular, or respiratory disease) or laboratory finding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters
  Parameters include: AUC, Cmax

SECONDARY OUTCOMES:
Safety and tolerability variables of fostamatinib 150mg: Adverse events, vital signs, physical examinations, clinical laboratory tests and electrocardiograms
Urine PK parameters of R406 and its N-glucuronide metabolite
  PK parameters including but not limited to Amount excreted (Ae) and renal clearance (CLr)
The effects of differences in protein binding by assessment of unbound R406 PK
  PK parameters including, but not limited to, unbound AUC and unbound Cmaxt

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, Study Director — AstraZeneca; Thomas Marbury, MD, Principal Investigator — Orlando Clinical
Locations (1):
- Research Site, Orlando, Florida, United States

REFERENCES:
- [Derived] Martin P, Oliver S, Gillen M, Marbury T, Millson D. Pharmacokinetic Properties of Fostamatinib in Patients With Renal or Hepatic Impairment: Results From 2 Phase I Clinical Studies. Clin Ther. 2015 Dec 1;37(12):2823-36. doi: 10.1016/j.clinthera.2015.09.016. Epub 2015 Oct 27. PMID 26519231
- See also: Related Info — http://www.studyforchange.com/